CLINICAL TRIAL: NCT04964713
Title: A Multicenter Clinical Study of Echocardiographic Assessment of Right Heart Function and Implications of Prognosis in Diabetes Mellitus
Brief Title: A Multicenter Clinical Study of Echocardiographic Assessment of Right Heart Function and Implications of Prognosis in Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Xie Mingxing (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shanghai Zhongshan Hospital (Other); Henan Provincial People's Hospital (Other); Wuhan Asia Heart Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xie Mingxing, Head of Department of Ultrasound, Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: 2021 V1.0
Record Dates: First submitted 2021-07-10; First posted 2021-07-16 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Prognosis
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- type 2 diabetes: T2DM was defined according to the WHO 2006 criteria. Assessing the left heart and right heart structure and function of T2DM by speckle tracking echocardiography.
- Prediabetes: According to the WHO 2006 criteria, combining impaired fasting glucose and impaired glucose tolerance as prediabetes. Assessing the left heart and right heart structure and function of prediabetes by speckle tracking echocardiography.
- normal glucose metabolism(NGM): Assessing the left heart and right heart structure and function of NGM by speckle tracking echocardiography.

SUMMARY:
The aims of this study are to 1. Evaluate the right heart structure and function in T2DM and Prediabetes patients by speckle tracking echocardiography, and to further investigate the influence of left heart on right heart structure and function in T2DM and Prediabetes patients. 2. To explore the prognostic value of right ventricular function in T2DM patients.

DETAILED DESCRIPTION:
This study will recruit 1000 T2DM patients and 500 Prediabetes and 500 healthy controls. Assessing the left heart and right heart structure and function by speckle tracking echocardiography. Patients with T2DM were followed up for adverse cardiovascular outcome events (myocardial infarction, cerebrovascular stroke, or cardiovascular death, hospitalization for heart failure). And the study aimed to 1. 1. Evaluate the right heart structure and function in T2DM and Prediabetes patients by speckle tracking echocardiography, and to further investigate the influence of left heart on right heart structure and function in T2DM and Prediabetes patients. 2. To explore the prognostic value of right ventricular function in T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

people with T2DM according to the WHO 2006 criteria

Exclusion Criteria:

including history or symptoms of CAD valvular heart disease, rhythm disturbances cardiomyopathy congenital heart disease symptomatic heart failure pulmonary disease

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with type 2 diabetes mellitus and prediabetes were diagnosed according to the WHO 2006 criteria, aged 35 -79 years, who are undergoing echocardiography examination in clinical needs.
Sampling Method: Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | through study completion, an average of 6 year
  including myocardial infarction, cerebrovascular stroke, or cardiovascular death, hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jing, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided